CLINICAL TRIAL: NCT03185910
Title: The Efficacy of a Mindfulness-Based Childbirth and Parenting Education on Pregnant Women's Childbirth Self-efficacy, Psychological Health and Maternal Outcomes: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Childbirth and Parenting Education on Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wan-Lin Pan, Nursing department, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104-E-20
Record Dates: First submitted 2017-05-27; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Stress, Psychological; Pregnancy Related
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCP education (Experimental): The intervention includes 3-hour classes per week during the duration of eight weeks and a 7- hour silent meditation practice as well.
  Interventions: Behavioral: MBCP education
- Hospital-based antenatal education (Placebo Comparator): Hospital-based antenatal education program will be held 2 hrs once a month for 2 months.
  Interventions: Behavioral: Hospital-based antenatal education

INTERVENTIONS:
Behavioral: MBCP education — MBCP education involves mindfulness breathing and other skills with mindfulness meditations.
  Arms: MBCP education
Behavioral: Hospital-based antenatal education — Hospital-based antenatal education involves all aspects of pregnancy, childbirth and postpartum.
  Arms: Hospital-based antenatal education

SUMMARY:
The purpose of this study is to explore the differences between stress, depression, childbirth self-efficacy, mindfulness and postnatal maternal outcomes in pregnant women with Mindfulness-Based Childbirth and Parenting education program.

DETAILED DESCRIPTION:
Being a mother is a huge change for women, and she will undergo a high degree of change and a strong threat in this transformation process. The purpose of this study is to explore the efficacy of a Mindfulness-Based Childbirth and Parenting(MBCP) Education Program on prenatal stress, depression, mindfulness, childbirth self-efficacy, and postnatal maternal outcomes.

Randomized Controlled Trial comparing two education programs with health and singleton pregnant women is run by the Random Allocation Software (Saghaei, 2004). Use the G-Power 3.1.9 windows: repeated measures and between factors among two groups to calculate the number of samples, and setting the power = .8, α = .05, effect size = .25. The estimated number of samples may be lost 20%, total 104 samples ( 52 samples in each group).

The protocol for the study used MBCP education, this program helps participants practice in the present moment, so that they may develop more confidence and well-being during pregnancy. The MBCP course is held for 3 hrs once a week for 8 weeks. They also had the home practice of 30 minutes a day with a DVD for the experimental group. The control group attending a hospital-based antenatal education program for 2 hrs once a month for 2 months from hospital staff nurses in all aspects of pregnancy, childbirth and postpartum. This study uses a standard verbal script to the eligible participants who were volunteers of pregnant women in the waiting room of metropolitan hospital in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were pregnant from 13th to 28th weeks gestation with a singleton pregnancy
* Subjects were at the age over 20
* Could speak and read Chinese fluently
* Willing and be able to attend the education program
* Determined to have a vaginal birth

Exclusion Criteria:

* Taking medication for diagnosing mental illness
* With complicated or high-risk pregnancies

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-12-02 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
change of prenatal and postnatal stress | Baseline, T1: After 2-month intervention, T2: At 36th week pregnancy, T3: 6 months after childbirth
  Self reported the perception of stress change from baseline to 6 months after childbirth using The Perceived Stress Scale

SECONDARY OUTCOMES:
postpartum medical records | After the childbirth within 24 hours will be collected
  This instrument was to explore whether recording of pregnancy outcome in medical records
change of symptoms with depression and anxiety | Baseline, T1: After 2-month intervention, T2: At 36th week pregnancy, T3: 6 months after childbirth
  Self reported the symptoms with depression and anxiety change from baseline to 6 months after childbirth using the Edinburgh Postnatal Depression Scale
change of the childbirth self-efficacy | Baseline, T1: After 2-month intervention, T2: At 36th week pregnancy, T3: 6 months after childbirth
  Self reported the childbirth self-efficacy change from baseline to 6 months after childbirth using the Childbirth Self-Efficacy Inventory
change of mindfulness | Baseline, T1: After 2-month intervention, T2: At 36th week pregnancy, T3: 6 months after childbirth
  Self reported the mindfulness change from baseline to 6 months after childbirth using Five Factor Mindfulness Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Lin Pan, MD, Principal Investigator — National Taipei University of Nursing and Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan WL, Chang CW, Chen SM, Gau ML. Assessing the effectiveness of mindfulness-based programs on mental health during pregnancy and early motherhood - a randomized control trial. BMC Pregnancy Childbirth. 2019 Oct 10;19(1):346. doi: 10.1186/s12884-019-2503-4. PMID 31601170